CLINICAL TRIAL: NCT02380118
Title: Intramuscular Olanzapine Versus Haloperidol or Midazolam for the Management of Acute Agitation in the Emergency Department - a Multicentre Randomised Clinical Trial
Brief Title: IM Olanzapine Versus Haloperidol or Midazolam
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary endpoint reached based on data projection from interim analysis.
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other); Tuen Mun Hospital (Other Government); Pamela Youde Nethersole Eastern Hospital (Other); Ruttonjee Hospital (Other); Prince of Wales Hospital, Shatin, Hong Kong (Other); United Christian Hospital (Other)
Responsible Party: Principal Investigator, Dr. Esther Wai Yin Chan, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PR/CT 0309/2014 (SC); HKU 789813M (Other Grant/Funding Number: Research Grant Council, Hong Kong)
Record Dates: First submitted 2015-01-29; First posted 2015-03-05 (Estimated); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Acute Agitation, Behavioural Emergency
Keywords: emergency; emergency medicine; sedation; acute agitation
MeSH Terms: conditions — Emergencies | interventions — Olanzapine; Haloperidol; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Olanzapine (Experimental): intramuscular olanzapine injection (zyprexa), 5 mg/dose, first dose and an optional second dose.
  Interventions: Drug: Olanzapine
- Haloperidol (Active Comparator): intramuscular haloperidol injection, 5 mg/dose, first dose and an optional second dose.
  Interventions: Drug: Haloperidol
- Midazolam (Active Comparator): intramuscular midazolam injection, 5 mg/dose, first dose and an optional second dose.
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Olanzapine — Intramuscular injection
  Other Names: ZYPREXA
  Arms: Olanzapine
Drug: Haloperidol — Intramuscular injection
  Arms: Haloperidol
Drug: Midazolam — Intramuscular injection
  Arms: Midazolam

SUMMARY:
The purpose of this study is to determine whether intramuscular olanzapine is safer (fewer adverse events) and more effective (shorter time to sedation) than conventional haloperidol or midazolam when used in the management of acute agitation in the emergency department.

DETAILED DESCRIPTION:
To address significant knowledge gaps by several means:

1. Investigate intramuscular use of sedative drugs within a predominantly Chinese population, to address this void in international literature impacting the management of acute agitation.

   The multi-centre RCT will determine the safety and efficacy of intramuscular olanzapine, in comparison with conventional medicines (haloperidol or midazolam) in a three-arm comparison for the sedation of acutely agitated patients in emergency department. Specifically, we aim to determine if administration of intramuscular olanzapine (a)is more effective than sedation with intramuscular haloperidol or intramuscular midazolam alone; (b)is safer than sedation with comparison arms; (c)decreases the amount of subsequent redosing or alternative drugs required; (d)is more favourable than the haloperidol and midazolam arms with respect to safety, efficacy and adverse events.
2. Investigate potential variables leading to emergency attendance and/or admission requiring parenteral sedation. These may include patient demographics and regular medications and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Emergency Department patients, requiring parenteral drug sedation (as determined by an emergency clinician) will be enrolled.

Exclusion Criteria:

* Patients will be excluded if there are

  1. known hypersensitivity or contraindication to the study drugs
  2. reversible aetiology for agitation (e.g. hypotension, hypoxia, hypoglycaemia)
  3. known pregnancy
  4. acute alcohol withdrawal
  5. patients aged>75 years.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Time to achieve adequate sedation | Within 60 minutes from drug administration
  Adequate sedation is determined by a 6-point validated scale.

SECONDARY OUTCOMES:
Total study drug doses administered; alternative drugs and doses used | From Emergency Department admission to transfer or discharge from AED, an expected average of 1 hour
Prolonged QTc interval | From Emergency Department admission to transfer or discharge from Emergency Department, an expected average of 1 hour
AED length of stay (LOS) | From Emergency Department admission to transfer or discharge from Emergency Department, an expected average of 1 hour
Adverse events | From Emergency Department admission to transfer or discharge from Emergency Department an expected average of 1 hour
  including airway management (jaw thrust, oral, nasal airway), need for assisted ventilation (bag/mask, intubation), oxygen desaturation <90%, systolic BP<90 mmHg, dystonic reactions, seizures, vomiting or aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Esther WY Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (6):
- Hong Kong (6):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Ruttonjee Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - United Christian Hospital, Hong Kong

REFERENCES:
- [Background] Knott JC, Bennett D, Rawet J, Taylor DM. Epidemiology of unarmed threats in the emergency department. Emerg Med Australas. 2005 Aug;17(4):351-8. doi: 10.1111/j.1742-6723.2005.00756.x. PMID 16091097
- [Background] Chan EW, Taylor DM, Knott JC, Phillips GA, Castle DJ, Kong DC. Intravenous droperidol or olanzapine as an adjunct to midazolam for the acutely agitated patient: a multicenter, randomized, double-blind, placebo-controlled clinical trial. Ann Emerg Med. 2013 Jan;61(1):72-81. doi: 10.1016/j.annemergmed.2012.07.118. Epub 2012 Sep 13. PMID 22981685
- [Background] Knott JC, Taylor DM, Castle DJ. Randomized clinical trial comparing intravenous midazolam and droperidol for sedation of the acutely agitated patient in the emergency department. Ann Emerg Med. 2006 Jan;47(1):61-7. doi: 10.1016/j.annemergmed.2005.07.003. Epub 2005 Aug 18. PMID 16387219
- [Background] Chan EW, Taylor DM, Knott JC, Kong DC. Variation in the management of hypothetical cases of acute agitation in Australasian emergency departments. Emerg Med Australas. 2011 Feb;23(1):23-32. doi: 10.1111/j.1742-6723.2010.01348.x. Epub 2010 Nov 22. PMID 21091874
- [Background] Chan EW, Knott JC, Taylor DM, Phillips GA, Kong DC. Intravenous olanzapine--another option for the acutely agitated patient? Emerg Med Australas. 2009 Jun;21(3):241-2. doi: 10.1111/j.1742-6723.2009.01190.x. No abstract available. PMID 19527287
- [Background] Chan EW, Taylor DM, Knott JC, Liew D, Kong DC. The pharmacoeconomics of managing acute agitation in the emergency department: what do we know and how do we approach it? Expert Rev Pharmacoecon Outcomes Res. 2012 Oct;12(5):589-95. doi: 10.1586/erp.12.53. PMID 23186399
- [Derived] Chan EW, Lao KSJ, Lam L, Tsui SH, Lui CT, Wong CP, Graham CA, Cheng CH, Chung TS, Lam HF, Ting SM, Knott JC, Taylor DM, Kong DCM, Leung LP, Wong ICK. Intramuscular midazolam, olanzapine, or haloperidol for the management of acute agitation: A multi-centre, double-blind, randomised clinical trial. EClinicalMedicine. 2021 Feb 11;32:100751. doi: 10.1016/j.eclinm.2021.100751. eCollection 2021 Feb. PMID 33681744